CLINICAL TRIAL: NCT03836053
Title: A Phase 1b Multicenter, Open-label, Expansion Study to Assess the Safety and Efficacy of AMG 420 as Monotherapy in Subjects With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Assessment of AMG 420 in Subjects With Relapsed and/or Refractory Multiple Myeloma
Acronym: AMG420
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Amgen re-evaluated the portfolio and decided to discontinue clinical development activities for AMG 420.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160370; 2018-002879-17 (EudraCT Number)
Record Dates: First submitted 2019-02-05; First posted 2019-02-11 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Phase 1b Primary objective Establish the safety and tolerability of AMG 420 at dose levels of 400 mcg/day and 600 mcg/day in subjects with relapsed and/or refractory multiple myeloma (RRMM)
  Phase 1b Key Secondary/Secondary objectives:
  Estimate overall response rate (ORR) and duration of response (DOR) Evaluate the rate of minimal residual disease (MRD)-negativity at the time of CR Establish the safety and tolerability of AMG 420 in subjects with extramedullary relapsed MM Characterize the PK of AMG 420 when administered as 4-week continuous IV infusion Evaluate other measures of anti-myeloma activity of AMG 420: Time to response, PFS, OS, TFI, BOR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMG 420 (Experimental): Single Arm Design
  Interventions: Drug: AMG 420

INTERVENTIONS:
Drug: AMG 420 — 28 day continuous Intravenous infusion of either 400 mcg/d or 600 mcg/d followed by 2 treatment free weeks

SUMMARY:
To confirm the maximum tolerated dose (MTD) from the BI 836909 trial of 400 mcg/d, given as 28-day continuous intravenous infusion in patients with relapsed and/or refractory multiple myeloma, to test the 600 mcg/d dose, given as a 28-day continuous iV infusion.

DETAILED DESCRIPTION:
Cohort 1 will consist of 10 subjects dosed at 400 mcg/d. Cohort 2 will consist of 10 subjects dosed at 600 mcg/d. All doses will be given as a 28-day continuous IV infusion, followed by a 2 week treatment-free interval, until subject experiences disease progression as per International Myeloma Working Group (IMWG) criteria.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject has provided informed consent prior to initiation of any study specific activities/procedures
2. Multiple myeloma meeting the following criteria:
3. Pathologically-documented diagnosis of multiple myeloma that is relapsed or is refractory as defined by the following: Relapsed after 3 or more lines of prior therapy that must include a proteasome inhibitors (PI), an immunomodulators (IMiD), and a CD38-directed monoclonal antibody in any order during the course of treatment OR refractory to a PI, IMiD, and CD38-directed monoclonal antibody.

   -Measurable disease, defined by 1 or more of the following at time of screening: 1) serum M-protein > 0.5 g/dL measured by serum protein electrophoresis (SPEP); 2) urinary M-protein excretion > 200 mg/24 hours; 3) Involved serum free light chain (sFLC ) measurement > 10 mg/dL, provided that the sFLC ratio is abnormal (<0.26 or >1.65) as per IMWG response criteria
4. . ECOG performance status of less than or equal to 2
5. Life expectancy of at least 3 months per PI judgement at screening
6. Hematological function without transfusion support (within 7 days from screening assessment) as follows:

   * ANC ≥ 1.0 x 10^9/L (without growth factor support)
   * platelet count ≥ 25 x 10^9/L (without transfusions)
   * hemoglobin ≥ 7.0 g/dL (transfusions permitted no later than 48 hours before screening)
7. Renal function as follows: calculated or measured creatinine clearance ≥30 mL/min using the Cockcroft-Gault equation or via 24-hour urine collection with plasma and urine creatinine concentrations, respectively
8. Hepatic function as follows: AST and ALT < 3x upper limit of normal (ULN); TBIL <1.5 x ULN (unless considered due to Gilbert's syndrome)

Key Exclusion Criteria:

1. Known central nervous system involvement by multiple myeloma
2. Evidence of primary or secondary plasma cell leukemia at the time of screening
3. Waldenstrom's macroglobulinemia
4. Unresolved toxicities from prior anticancer therapy, defined as not having resolved to CTCAE version 5.0 grade 1 or to levels dictated in the eligibility criteria with the exception of grade 2 peripheral neuropathy, alopecia, or toxicities from prior anticancer therapy that are considered irreversible (defined as having been present and stable for > 4 weeks) which may be allowed if they are not otherwise described in the exclusion criteria and there is agreement to allow by the PI and Amgen medical monitor
5. History of other malignancy within the past 3 years, with the following exceptions: 1. malignancy treated with curative intent and with no known active disease present for ≥ 1 year before enrollment and felt to be at low risk for recurrence by the treating physician; 2. adequately-treated non-melanoma skin cancer or lentigo maligna without evidence of disease; 3. adequately-treated cervical carcinoma in situ without evidence of disease; 4. breast ductal carcinoma in situ with full surgical resection (ie, negative margins) and without evidence of disease; 5. prostate cancer with a Gleason score < 6 with undetectable PSA over 12 months; 6. treated medullary or papillary thyroid cancer; 7. adequately-treated urothelial papillary noninvasive carcinoma or carcinoma in situ; similar neoplastic conditions with an expectation of > 95% five-year disease-free survival; 8. see exclusion criterion # 2 for exclusion of subjects with evidence of primary or secondary plasma cell leukemia at the time of screening
6. Known history of amyloidosis
7. Current or known history of autoimmune diseases requiring systemic treatment in past 5 years except vitiligo, resolved childhood asthma/atopy, or subjects with history of hypothyroidism after completing treatment for autoimmune thyroid disease, stable on hormone replacement therapy.
8. Clinically not-controlled chronic or ongoing infectious disease requiring treatment at the time of study day 1 or within the 14 days before study day 1
9. Symptomatic peripheral sensory or motor neuropathy of grade ≥3
10. History or presence of clinically relevant central nervous system (CNS) pathology as uncontrolled epilepsy or seizure disorder, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, and psychosis
11. Active hepatitis B and C based on the following results: a) Positive for HepBsAg; b) Negative HepBsAg and positive for hepatitis B core antibody; c) Positive Hepatitis C virus antibody (HepCAb)
12. Known or suspected HIV infection or subjects who are HIV seropositive
13. Baseline ECG QTc > 470 msec (applying Fridericia correction)
14. Previously received an allogeneic stem cell transplant and the occurrence of 1 or more of the following: a) received the transplant within 6 months prior to study day 1; b) received immunosuppressive therapy within the last 3 months prior to study day 1; c) any active acute graft versus host disease (GvHD), grade 2 to 4, according to the Glucksberg criteria or active chronic GvHD requiring systemic treatment; d) any systemic therapy against GvHD within 2 weeks prior to start of investigational product treatment
15. Autologous stem cell transplantation < 90 days prior to study day 1
16. Treatment with systemic immune modulators including, but not limited to, nontopical systemic corticosteroids (unless the dose is ≤ 10 mg/day prednisone or equivalent), cyclosporine, and tacrolimus within 2 weeks before study day 1
17. Last anticancer treatment < 2 weeks prior to study day 1
18. Last treatment with a therapeutic antibody less than 4 weeks prior to study day 1
19. Systemic radiation therapy within 28 days prior to study day 1. Focal radiotherapy within 14 days prior to study day 1.
20. Major surgery defined as surgery requiring general anesthesia with endotracheal intubation within 28 days prior to study day 1, unless discussed with and eligibility approved by Amgen medical monitor
21. Prior treatment with any drug that specifically targets BCMA on tumor cells (eg, other bi-specific antibody constructs, antibody drug conjugates, or CAR T-cells, except for subjects who were previously treated with AMG 420 in this study and who are candidates for second-course treatment
22. Treatment with medications known to cause QTc interval prolongation within the washout periods described in Section 12.10 unless approved by the Amgen medical monitor
23. Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
24. History or evidence of any other clinically-significant disorder, condition, or disease (eg, symptomatic congestive heart failure, unstable angina pectoris,cardiac arrhythmia requiring therapy at time of screening) with the exception of those outlined above that, in the opinion of the investigator or Amgen medical monitor, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (10):
- United States (4):
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
- Australia (2):
  - St Vincents Hospital Sydney, Darlinghurst, New South Wales
  - St Vincents Hospital Melbourne, Fitzroy, VIC, Victoria
- Belgium (2):
  - Centres Hospitaliers Jolimont - Hopital de Jolimont, Haine Saint Paul - La Louviere
  - Centre Hospitalier Universitaire Dinant Godinne - Universite Catholique de Louvain Namur, Yvoir
- National Hospital Organization Okayama Medical Center, Okayama, Okayama-ken, Japan
- Kantonsspital St Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Rodriguez C, Rodriguez T, Kentos A, Driessen C, Sunami K, Lesokhin AM, Yee AJ, Minella AC, Maraboina R, Upreti VV, Zhou D, Shabooti M, Stieglmaier J, Quach H. BCMA-targeting BiTE molecule AMG 420 in relapsed or refractory multiple myeloma: a phase 1b open-label expansion study. Leuk Lymphoma. 2025 Nov;66(11):2108-2117. doi: 10.1080/10428194.2025.2528115. Epub 2025 Jul 21. PMID 40690374
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 10 centers in Australia, Belgium, Japan, Switzerland, and the United States from 04 March 2019 to 21 April 2022.
Pre-assignment Details: 23 participants were enrolled and all 23 of those participants received study drug.
Groups:
- AMG 420 200 µg/Day: 28 day continuous intravenous infusion of AMG 420 200 µg/day followed by a 2 week treatment-free interval, until progressive disease (PD) or relapse as defined by International Myeloma Working Group (IMWG) response criteria, unacceptable safety events, next anti-multiple myeloma treatment, or other reason for permanent treatment discontinuation
- AMG 420 400 µg/Day: 28 day continuous intravenous infusion of AMG 420 400 µg/day followed by a 2 week treatment-free interval, until PD or relapse as defined by IMWG response criteria, unacceptable safety events, next anti-multiple myeloma treatment, or other reason for permanent treatment discontinuation
- AMG 420 600 µg/Day: 28 day continuous intravenous infusion of AMG 420 600 µg/day followed by a 2 week treatment-free interval, until PD or relapse as defined by IMWG response criteria, unacceptable safety events, next anti-multiple myeloma treatment, or other reason for permanent treatment discontinuation
Period: Overall Study
Arm/Group | AMG 420 200 µg/Day | AMG 420 400 µg/Day | AMG 420 600 µg/Day
Started | 1 | 12 | 10
Completed | 0 | 2 | 0
Not Completed | 1 | 10 | 10
Not completed — Protocol-specified criteria | 0 | 2 | 1
Not completed — Death | 1 | 6 | 4
Not completed — Withdrawal of consent from study | 0 | 0 | 1
Not completed — Decision by sponsor | 0 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Safety analysis set includes all participants who enrolled and received at least 1 dose of AMG 420.
Groups:
- Total: Total of all reporting groups
Arm/Group | AMG 420 200 µg/Day | AMG 420 400 µg/Day | AMG 420 600 µg/Day | Total
Number analyzed (Participants) | 1 | 12 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (NA) — NA because there was only 1 participant analyzed. | 64.7 (6.7) | 60.8 (11.7) | 62.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 5 | 9
  Male | 0 | 9 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 12 | 10 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 3 | 5
  White | 0 | 10 | 7 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLTs were graded using Common Terminology Criteria for Adverse Events (CTCAE) v5.0, with the exception of cytokine release syndrome (CRS) and tumor lysis syndrome (TLS), which graded using the criteria referenced in the publication by Lee et al, 2014 and the Cairo Bishop criteria referenced in the publication by Coiffier et al, 2008 respectively.
  A participant was non-DLT evaluable if they dropped out before completion of the DLT-evaluable period for reasons other than a DLT.
Time Frame: Day 1 to Week 4
Population: DLT evaluation analysis set includes participants who completed the DLT evaluable period or experienced a DLT any time during the DLT evaluable period.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 420 200 µg/Day | AMG 420 400 µg/Day | AMG 420 600 µg/Day
Number analyzed (Participants) | 1 | 11 | 8
Participants | 1 | 1 | 0

2. Primary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: The severity of TEAEs were graded using the CTCAE version 5.0 with the exception of CRS and TLS, which graded using the criteria referenced in the publication by Lee et al, 2014 and the Cairo Bishop criteria referenced in the publication by Coiffier et al, 2008. Any clinically significant changes in vital signs, electrocardiograms (ECGs) and clinical laboratory tests were recorded as TEAEs.
Time Frame: Up to approximately 3 years
Population: Safety analysis set defined as all participants that are enrolled and receive at least 1 dose of AMG 420.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 420 200 µg/Day | AMG 420 400 µg/Day | AMG 420 600 µg/Day
Number analyzed (Participants) | 1 | 12 | 10
Participants | 1 | 12 | 10

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants for whom the best overall response was a stringent complete response (CR), CR, very good partial response (PR), or partial response as determined by the IMWG Uniform Response Criteria. The ORR along with the associated 95% exact binomial confidence interval (Clopper Pearson Method) was determined.
Time Frame: Up to approximately 3 years
Population: Safety analysis set includes all participants who enrolled and received at least 1 dose of AMG 420.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AMG 420 200 µg/Day | AMG 420 400 µg/Day | AMG 420 600 µg/Day
Number analyzed (Participants) | 1 | 12 | 10
Percentage of participants | 0 [0.00 to 97.50] | 41.7 [15.17 to 72.33] | 30.0 [6.67 to 65.25]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as number of months between first objective response to progressive disease or death (due to any cause), whichever occurred first.
  Kaplan-Meier methods were used to estimate the distribution of DOR. The median and corresponding two-sided 95% confidence intervals were calculated.
Time Frame: Up to approximately 3 years
Population: Safety analysis set includes all participants who enrolled and received at least 1 dose of AMG 420.
  DOR was only calculated for participants who experienced a best overall response of partial response or better.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AMG 420 200 µg/Day | AMG 420 400 µg/Day | AMG 420 600 µg/Day
Number analyzed (Participants) | 0 | 5 | 3
Months |  | 5.49 [1.41 to NA] — Not enough responses to calculate upper limit of 95% CI | NA [1.45 to NA] — Not enough responses to calculate a median or upper limit of 95% CI

5. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD) Negativity Response at CR
Description: MRD negativity at CR or better assessed by using the IMWG criteria.
  Percentage of MRD negative responders at CR along with exact 2- sided 95% were provided by using the Clopper Pearson method.
Time Frame: Up to approximately 3 years
Population: Safety analysis set includes all participants who enrolled and received at least 1 dose of AMG 420.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AMG 420 200 µg/Day | AMG 420 400 µg/Day | AMG 420 600 µg/Day
Number analyzed (Participants) | 1 | 12 | 10
Percentage of participants | 0.0 [0.0 to 97.50] | 8.3 [0.21 to 38.48] | 10.0 [0.25 to 44.50]

6. Primary Outcome: Number of Participants Who Experienced a Treatment-related TEAE
Description: The severity of treatment-related TEAEs were graded using the CTCAE version 5.0 with the exception of CRS and TLS, which graded using the criteria referenced in the publication by Lee et al, 2014 and the Cairo Bishop criteria referenced in the publication by Coiffier et al, 2008.
  Treatment-related TEAEs were those that were considered related to the study treatment by the investigator.
Time Frame: Up to approximately 3 years
Population: Safety analysis set defined as all participants that are enrolled and receive at least 1 dose of AMG 420.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 420 200 µg/Day | AMG 420 400 µg/Day | AMG 420 600 µg/Day
Number analyzed (Participants) | 1 | 12 | 10
Participants | 1 | 12 | 9

7. Secondary Outcome: Number of Participants With Minimal Residual Disease (MRD) Negativity Response at CR
Description: Number of participants with MRD negativity at CR or better assessed by using the IMWG criteria.
Time Frame: Up to approximately 3 years
Population: Safety analysis set includes all participants who enrolled and received at least 1 dose of AMG 420.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 420 200 µg/Day | AMG 420 400 µg/Day | AMG 420 600 µg/Day
Number analyzed (Participants) | 1 | 12 | 10
Participants | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Up to approximately 3 years
Description: Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug. All-cause mortality is reported for all participants enrolled in the study.
Groups:
- Total: AMG 420 Total
Arm/Group | AMG 420 200 µg/Day | AMG 420 400 µg/Day | AMG 420 600 µg/Day | Total
All-Cause Mortality (participants affected / at risk) | 1/1 | 6/12 | 4/10 | 11/23
Serious Adverse Events (participants affected / at risk) | 1/1 | 10/12 | 8/10 | 19/23
Other Adverse Events (participants affected / at risk) | 1/1 | 12/12 | 10/10 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 420 200 µg/Day (N=1) | AMG 420 400 µg/Day (N=12) | AMG 420 600 µg/Day (N=10) | Total (N=23)
Asthenia (General disorders) | 0 | 1 | 0 | 1
Disease progression (General disorders) | 0 | 2 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 2 | 2
Cytokine release syndrome (Immune system disorders) | 0 | 5 | 3 | 8
Bacteraemia (Infections and infestations) | 0 | 1 | 1 | 2
Device related infection (Infections and infestations) | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 1
Infusion site infection (Infections and infestations) | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 1 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 3
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 420 200 µg/Day (N=1) | AMG 420 400 µg/Day (N=12) | AMG 420 600 µg/Day (N=10) | Total (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 | 4 | 4 | 8
Hyperfibrinogenaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Leukocyte vacuolisation (Blood and lymphatic system disorders) | 0 | 0 | 2 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 5
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1 | 2
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 1
Diplopia (Eye disorders) | 0 | 1 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 3 | 5 | 8
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 5 | 3 | 8
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Chest discomfort (General disorders) | 0 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 5 | 6 | 11
Hypothermia (General disorders) | 0 | 0 | 1 | 1
Malaise (General disorders) | 0 | 1 | 0 | 1
Oedema (General disorders) | 0 | 2 | 0 | 2
Oedema peripheral (General disorders) | 0 | 2 | 3 | 5
Peripheral swelling (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 6 | 6 | 12
Ulcer (General disorders) | 0 | 0 | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 9 | 7 | 17
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 1
Metapneumovirus infection (Infections and infestations) | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 2 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1 | 2 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 4 | 1 | 5
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 1
Blood creatine increased (Investigations) | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1
Blood fibrinogen increased (Investigations) | 0 | 0 | 1 | 1
C-reactive protein increased (Investigations) | 0 | 1 | 1 | 2
Carbon dioxide decreased (Investigations) | 0 | 0 | 1 | 1
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 1 | 2
Fibrin D dimer increased (Investigations) | 0 | 0 | 2 | 2
Immature granulocyte count increased (Investigations) | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1
Nitrite urine present (Investigations) | 0 | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 2 | 1 | 3
Protein total increased (Investigations) | 0 | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 2 | 2 | 4
Weight increased (Investigations) | 0 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 1 | 2
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 4 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 4 | 6
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 4
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 3 | 5
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 8 | 4 | 12
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 1 | 1 | 2
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1
Nervousness (Psychiatric disorders) | 0 | 1 | 0 | 1
Substance abuse (Psychiatric disorders) | 0 | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 3
Hypertension (Vascular disorders) | 0 | 1 | 1 | 2
Hypotension (Vascular disorders) | 0 | 1 | 2 | 3

LIMITATIONS AND CAVEATS:
The study was terminated early due to sponsor decision and long-term follow-up was cancelled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT03836053/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT03836053/SAP_001.pdf